CLINICAL TRIAL: NCT03566979
Title: A Randomized, Double-Blind, Placebo- and Active- Controlled, Efficacy and Safety Study of a Test Naproxen Sodium 220 mg Tablet in Postoperative Dental Pain
Brief Title: Efficacy and Safety Study of a Test Naproxen Sodium 220mg Tablet in Postoperative Dental Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc., McNeil Consumer Healthcare Division (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCSPAA000457
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Results first posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Post-operative Dental Pain

STUDY DESIGN:
Intervention Model Description: Post-operative dental pain following third molar extraction.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Test naproxen sodium tablet (Experimental): Single dose of 440 mg of naproxen sodium administered as two Test Naproxen Sodium 220 mg tablets (Test NPX)
  Interventions: Drug: Test naproxen sodium tablet
- Commercial naproxen sodium tablet (Active Comparator): Single dose of 440 mg of naproxen sodium administered as two commercial naproxen sodium 220 mg tablets
  Interventions: Drug: Commercial naproxen sodium tablet
- Commercial naproxen sodium liquid gels capsule (Active Comparator): Single dose of 440 mg of naproxen sodium administered as two 220 mg commercial liquid gels capsules
  Interventions: Drug: Commercial naproxen sodium liquid gels capsule
- Placebo tablet (Placebo Comparator): Single dose of two Placebo tablets
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: Test naproxen sodium tablet — Single dose of 2 test naproxen sodium 220 mg tablets
  Other Names: Test NPX tablet
  Arms: Test naproxen sodium tablet
Drug: Commercial naproxen sodium tablet — Single dose of 2 naproxen sodium 220 mg tablets
  Other Names: Commercial NPX tablet
  Arms: Commercial naproxen sodium tablet
Drug: Commercial naproxen sodium liquid gels capsule — Single dose of 2 naproxen sodium 220 mg liquid gel capsules
  Other Names: Commercial NPX liquid gels capsule
  Arms: Commercial naproxen sodium liquid gels capsule
Drug: Placebo tablet — 2 placebo tablets
  Arms: Placebo tablet

SUMMARY:
To evaluate analgesic onset, efficacy, and safety of a single dose of 440 mg of naproxen sodium administered as two Test Naproxen Sodium 220 mg tablets compared with two commercial naproxen sodium products (two naproxen sodium 220 mg tablets and two naproxen sodium 220 mg liquid gels capsules) and placebo in the dental pain model following third-molar extractions.

DETAILED DESCRIPTION:
This is a single-dose, randomized, double-blind, placebo- and active- controlled, parallel-group study to evaluate the analgesic onset, efficacy, and safety profile of 440 mg of naproxen sodium administered as two Test NPX 220 mg tablets compared with two commercial products and placebo over a twelve-hour period after third-molar extractions. Subjects will undergo dental extraction of three or four third molars.

ELIGIBILITY:
Inclusion Criteria:

1. 17 - 50 years old
2. Weigh 100 pounds or greater and have a body mass index (BMI) of 17.5 to 30.4 (inclusive) at screening
3. Dental extraction of three or four third molars
4. Meets post-surgical pain
5. Females of childbearing potential and males agree to contraceptive requirements of study
6. Have a negative urine drug screen at screening, and on day of surgical procedure

Exclusion Criteria:

1. Pregnant female, breastfeeding, trying to be pregnant or male with pregnant partner or partner currently trying to become pregnant
2. Have a known allergy or hypersensitivity to naproxen or other NSAIDs, including aspirin, or to acetaminophen, hydrocodone or other opioids
3. Not able to swallow large tablets or capsules
4. History of any condition (s) in investigator's opinion, may jeopardize subject safety, well-being and integrity of study
5. Use analgesics 5 or more times per week
6. History of chronic tranquilizer use, heavy drinking, substance abuse as judged by investigator site staff within last 5 years
7. Use of immunosuppressive drugs within 2 weeks of screening
8. History of endoscopically documented peptic ulcer disease or bleeding disorder in last 2 years

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 501 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Bertoch, MD, Principal Investigator — JBR Clinical Research
Locations (1):
- JBR Clinical Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Single dose of two Placebo tablets.
- Test Naproxen Sodium 440 Milligram (mg): Single dose of 440 mg of naproxen sodium administered as two Test Naproxen Sodium 220 mg tablets (Test NPX).
- Commercial Naproxen Sodium Tablet 440 mg: Single dose of 440 mg of naproxen sodium administered as two commercial naproxen sodium 220 mg tablets.
- Commercial Naproxen Sodium Liquid Gel Capsule 440 mg: Single dose of 440 mg of naproxen sodium administered as two 220 mg commercial liquid gels capsules.
Period: Overall Study
Arm/Group | Placebo | Test Naproxen Sodium 440 Milligram (mg) | Commercial Naproxen Sodium Tablet 440 mg | Commercial Naproxen Sodium Liquid Gel Capsule 440 mg
Started | 58 | 152 | 142 | 149
Completed | 53 | 145 | 132 | 143
Not Completed | 5 | 7 | 10 | 6
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 1
Not completed — Lost to Follow-up | 2 | 7 | 9 | 5
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported in all randomized participants who have received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Test Naproxen Sodium 440 Milligram (mg) | Commercial Naproxen Sodium Tablet 440 mg | Commercial Naproxen Sodium Liquid Gel Capsule 440 mg | Total
Number analyzed (Participants) | 58 | 152 | 142 | 149 | 501
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.1 (2.11) | 18.9 (2.2) | 18.9 (2.34) | 19.1 (2.3) | 19 (2.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 81 | 77 | 75 | 262
  Male | 29 | 71 | 65 | 74 | 239
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 20 | 20 | 20 | 71
  Not Hispanic or Latino | 46 | 132 | 121 | 129 | 428
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 2 | 5
  Asian | 0 | 3 | 3 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 0 | 2
  Black or African American | 2 | 1 | 2 | 3 | 8
  White | 51 | 140 | 126 | 134 | 451
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 9 | 5 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58 | 152 | 142 | 149 | 501

OUTCOME MEASURES:

1. Primary Outcome: Time to Confirmed Perceptible Pain Relief
Description: Minutes until confirmed first perceptible pain relief was achieved. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The first perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief.
Time Frame: 12 hours
Population: Population analyzed included all randomized participants.
Measure: Median (Full Range); unit: Minutes
Groups:
- Test Naproxen Sodium Tablet (440 mg): Single dose of 440 mg of naproxen sodium administered as two Test Naproxen Sodium 220 mg tablets (Test NPX).
- Commercial Naproxen Sodium Tablets (440 mg): Single dose of 440 mg of naproxen sodium administered as two commercial naproxen sodium 220 mg tablets.
- Commercial Naproxen Sodium Liquid Gel Capsules (440 mg): Single dose of 440 mg of naproxen sodium administered as two 220 mg commercial liquid gels capsules.
Arm/Group | Placebo | Test Naproxen Sodium Tablet (440 mg) | Commercial Naproxen Sodium Tablets (440 mg) | Commercial Naproxen Sodium Liquid Gel Capsules (440 mg)
Number analyzed (Participants) | 58 | 152 | 142 | 149
Minutes | NA [3 to 720] — Here NA signifies that median is not estimable as less than 50% of the participants obtained confirmed perceptible pain relief by 12 hours. | 18.7 [2 to 720] | 23.5 [2.5 to 720] | 28.1 [2.1 to 720]

2. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Pain Relief From 45 Minutes to Successively Earlier Minutes in One-minute Increments
Description: Percentage of participants with confirmed perceptible pain relief from 45 minutes to successively earlier minutes in one-minute increments were reported.
Time Frame: Up to 45 minutes after dosing
Population: Population analyzed included all randomized participants. Data for this outcome measure was planned to be analyzed and reported only for Placebo and Test NPX (440 mg) arms.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test Naproxen Sodium Tablet (440 mg)
Number analyzed (Participants) | 58 | 152
Percentage of Participants
  45 minutes after dosing | 27.6 | 84.9
  44 minutes after dosing | 25.9 | 84.9
  43 minutes after dosing | 25.9 | 84.2
  42 minutes after dosing | 25.9 | 84.2
  41 minutes after dosing | 25.9 | 84.2
  40 minutes after dosing | 25.9 | 84.2
  39 minutes after dosing | 25.9 | 84.2
  38 minutes after dosing | 25.9 | 84.2
  37 minutes after dosing | 24.1 | 84.2
  36 minutes after dosing | 24.1 | 84.2
  35 minutes after dosing | 24.1 | 83.6
  34 minutes after dosing | 24.1 | 82.9
  33 minutes after dosing | 24.1 | 82.2
  32 minutes after dosing | 22.4 | 81.6
  31 minutes after dosing | 20.7 | 80.3
  30 minutes after dosing | 20.7 | 74.3
  29 minutes after dosing | 19.0 | 71.7
  28 minutes after dosing | 19.0 | 69.1
  27 minutes after dosing | 19.0 | 69.1
  26 minutes after dosing | 19.0 | 67.8
  25 minutes after dosing | 17.2 | 67.8
  24 minutes after dosing | 17.2 | 65.8
  23 minutes after dosing | 17.2 | 63.2
  22 minutes after dosing | 17.2 | 61.8
  21 minutes after dosing | 17.2 | 57.9
  20 minutes after dosing | 17.2 | 53.9
  19 minutes after dosing | 17.2 | 50.7
  18 minutes after dosing | 17.2 | 47.4
  17 minutes after dosing | 17.2 | 45.4
  16 minutes after dosing | 12.1 | 42.1
  15 minutes after dosing | 12.1 | 32.2
  14 minutes after dosing | 8.6 | 23.0
  13 minutes after dosing | 8.6 | 17.1

ADVERSE EVENTS:
Time Frame: Up to Day 70
Description: The safety analysis dataset included all participants who took at least one dose of study medication and had any follow-up information.
Arm/Group | Placebo | Test Naproxen Sodium 440 Milligram (mg) | Commercial Naproxen Sodium Tablet 440 mg | Commercial Naproxen Sodium Liquid Gel Capsule 440 mg
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/152 | 0/142 | 0/149
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/152 | 0/142 | 0/149
Other Adverse Events (participants affected / at risk) | 6/58 | 2/152 | 6/142 | 4/149
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=58) | Test Naproxen Sodium 440 Milligram (mg) (N=152) | Commercial Naproxen Sodium Tablet 440 mg (N=142) | Commercial Naproxen Sodium Liquid Gel Capsule 440 mg (N=149)
Nausea (Gastrointestinal disorders) | 6 | 0 | 5 | 2
Vomiting (Gastrointestinal disorders) | 3 | 2 | 2 | 3

LIMITATIONS AND CAVEATS:
No study limitation was reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT03566979/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT03566979/SAP_001.pdf